CLINICAL TRIAL: NCT01777269
Title: A Prospective Study of Sexual Function in Sexually Active Men Treated for BPH
Brief Title: Prospective Sexual Function Study for BPH Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116115; 2012-002047-26 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duodart (Experimental): Fixed dose combination of dutasteride 0.5mg and tamsulosin 0.4mg. A capsule once daily during 12 months
  Interventions: Drug: Dutasteride plus tamsulosin
- Sugar Pill (Placebo Comparator): A capsule once daily during 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride plus tamsulosin — Take 1 capsule daily
  Arms: Duodart
Drug: Placebo — Take one capsule daily
  Arms: Sugar Pill

SUMMARY:
This is an European double-blind, placebo controlled parallel group comparison of DUODART (fixed dose combination of dutasteride 0.5mg and tamsulosin 0.4mg, one capsule daily) and placebo.

PRIMARY OBJECTIVE:

To assess the change in sexual function from baseline to 1 year in sexually active men with at least moderate BPH who are treated with DUODART, compared to men treated with placebo .

DETAILED DESCRIPTION:
This is an European double-blind, placebo controlled parallel group comparison of DUODART (fixed dose combination of dutasteride 0.5mg and tamsulosin 0.4mg, one capsule daily) and placebo. Men eligible at screening will be randomised, after a 4 week placebo run-in, to the 2 treatment groups in a 1:1 ratio. All men will receive standardised lifestyle advice (primarily concerning weight management and exercise) relevant to maintaining sexual function. Men will also receive a standardised lifestyle advice leaflet for BPH. The double blind phase will continue for 12 months, with assessment visits at 2 weeks and at months 1, 3, 6, 9 and a final visit at month 12. Subjects with sexual adverse events during the double blind phase will continue to be followed at scheduled study visits until resolution of the adverse event or at a visit 6 months after the last dose of study medication, whichever is sooner.

PRIMARY OBJECTIVE:

To assess the change in sexual function from baseline to 1 year in sexually active men with at least moderate BPH (international prostate symptom score - IPSS = or > 12) who are treated with DUODART, compared to men treated with placebo . Change in sexual function will be assessed by change in total score from the full men's sexual health questionnaire (MSHQ) which has domains for erectile dysfunction, ejaculatory function and libido.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥50 years.
* Men must be sexually active. A man is considered sexually active if he has been engaged in sexual activity with a partner during the past 4 weeks (at least once) and plans to be active during the next 4 weeks (unless due to travel or other practical reasons). Men should confirm that they are in a stable relationship and expect to maintain their sexual activity over the next year.
* A confirmed clinical diagnosis of BPH.
* International Prostate Symptom Score (IPSS) ≥12 at Visit 1 (screening), with bother score 4 or less (score from the IPSS Quality of Life question 8).
* Prostate volume ≥30 cc (by transrectal ultrasonography; TRUS). Measurement should be available by the baseline visit and should have been made /arranged at the screening visit or within the previous 6 months.
* Total serum prostate specific antigen (PSA ≥1.5 ng/mL (see exclusion criteria 1) at Visit 1 (screening).
* Willing and able to give signed written informed consent and comply with study procedures, including the ability to participate in the study for the full 1 year (or 18 months if necessary because of a persistent sexual AE).
* Fluent and literate in local language with the ability to read, comprehend and record information on the MSHQ, IPSS, PPSM, BPH Impact Index (BII) and C-SSRS questionnaires.
* Able to swallow and retain oral medication.
* Men with a female partner of childbearing potential must either agree to use effective contraception or have had a prior vasectomy. Contraception must be used from 2 weeks prior to administration of the first dose of study treatment until at least 5 half-lives for the drug (45 days) plus 3 months (i.e. a total of 4.5 months) to allow clearance of any altered sperm after the last dose of study treatment.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Total serum PSA >10.0 ng/mL at Visit 1 (screening).
* History or evidence of prostate cancer (e.g. positive biopsy or ultrasound, suspicious DRE and/or rising PSA). Subjects with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable PSA are eligible for the study.

Note: If total serum PSA is >4ng/mL and unless PSA value has been stable for at least the past 2 years, the investigator should make every appropriate effort to exclude the possibility of prostate cancer, including consideration of prostate biopsy.

Excluded medication and therapies

* Current or prior use (within the periods given) of the following prohibited medications
* Any prior use of a 5α-reductase inhibitor (finasteride or dutasteride),
* Anti-cholinergics (e.g. oxybutynin, propantheline, tolerodine, solifenacin or darifenacin) within 1 month prior to visit 2 (baseline)
* An alpha-adrenoreceptor blocker (i.e. indoramin, prazosin, terazosin, tamsulosin, alfuzosin and doxazosin) within 1 month prior to visit 2 (baseline)
* Use of any drugs with anti-androgenic properties (e.g. spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, progestational agents) within the 6 months prior to visit 1 (screening).
* Use of any drugs noted for propensity to cause gynaecomastia, or which could affect prostate volume, within 6 months prior to Visit 1 (screening).
* Use of any investigational or marketed study drug within 30 days or 5 half-lives of the drug in question, (whichever is longer), preceding visit 2 (baseline).
* Current use (at the baseline visit or within the prior 1month) of:
* PDE-5 inhibitors for Erectile Dysfunction.
* Anabolic steroids.
* Drugs known or thought to have an interaction with tamsulosin, e.g. cimetidine and warfarin.
* Use of phytotherapy for BPH within 2 weeks prior to Visit 1 (screening) and/or predicted to need phytotherapy during the study.
* History of a known (immediate or delayed) hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to the study medication or excipients that, in the opinion of the Investigator or GSK, contraindicate their participation.
* Previous prostatic surgery (including TURP, balloon dilatation, thermotherapy and stent replacement) or other invasive or minimally invasive procedures to treat BPH.

Recent Medical Procedures

- History of flexible/rigid cystoscopy or other instrumentation of the urethra within 7 days prior to Visit 1 (screening). Catheterisation (<10F) is acceptable with no time restriction.

Medical history

* Presence of structural abnormalities in the Lower Urinary Tract or sexual organs (e.g. urethral stricture, Peyronie's Disease etc) that may cause LUTS or sexual dysfunction.
* History of AUR.
* Post-void residual volume >100 mL (suprapubic ultrasound) at Visit 1 (screening) or a recorded PVR above this level on any previous examination. Measurement should be available by the baseline visit and should have been made /arranged at the screening visit or within the previous 6 months.
* Any causes other than BPH, which may in the judgement of the investigator, result in urinary symptoms (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, or acute or chronic urinary tract infections).
* History of 'first dose' hypotensive episode on initiation of alpha-1-adrenoreceptor antagonist therapy.
* History of postural hypotension, dizziness, vertigo or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* History of breast cancer or clinical breast examination finding of unclear origin or suggestive of malignancy.
* Prior history of malignancies (other than basal cell carcinoma or squamous cell carcinoma of the skin) within the past 5 years. Subjects with an earlier history of malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* History of hepatic impairment or abnormal liver function tests at Visit 1 (screening) (defined as ALT, AST or alkaline phosphatase >2 times the ULN, or total bilirubin >1.5 times the ULN (unless associated with predominantly indirect bilirubin elevation or Gilbert's syndrome).
* History of renal insufficiency, or serum creatinine >1.5 times the upper limit of normal at Visit 1 (screening).
* Any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to the Screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History or current evidence of drug or alcohol abuse within the previous 12 months.
* History or presence of any serious and/or unstable pre-existing psychiatric disorder or other conditions that in the opinion of the Investigator or GSK Medical Monitor, could interfere with subject's safety, obtaining informed consent, compliance to the study procedures, or confound the results of the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (59):
- Australia (8):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Wahroonga, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Malvern, Victoria
- France (6):
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Thouars
- Germany (15):
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Strausberg, Brandenburg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Buchholz, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Dülmen, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Wedel, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Eisleben Lutherstadt
- Greece (3):
  - GSK Investigational Site, Argos
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Larissa
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Szentes
- Netherlands (8):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Doetinchem
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Winterswijk
- Spain (14):
  - GSK Investigational Site, Alcazar de San Juan (Ciudad Real)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bormujo (Sevilla)
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Coslada
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Mendaro, Guipuzcoa
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Toledo
  - GSK Investigational Site, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Roehrborn CG, Manyak MJ, Palacios-Moreno JM, Wilson TH, Roos EPM, Santos JC, Karanastasis D, Plastino J, Giuliano F, Rosen RC. A prospective randomised placebo-controlled study of the impact of dutasteride/tamsulosin combination therapy on sexual function domains in sexually active men with lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH). BJU Int. 2018 Apr;121(4):647-658. doi: 10.1111/bju.14057. Epub 2017 Nov 16. PMID 29044968
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a European double-blind, placebo-controlled, parallel-group study to assess the impact of dutasteride treatment on sexual function in men with moderate/severe Benign Prostatic Hyperplasia (BPH)
Pre-assignment Details: Eligible participants (par.) entered a 4-week Placebo Run-in Phase, and were randomised in 1:1 ratio to receive DUODART (fixed dose combination of dutasteride 0.5 mg and tamsulosin 0.4 mg) and placebo one capsule daily for 52 weeks. Follow-up was performed 6 months after the last dose of study medication
Groups:
- Placebo: Participants received a matching placebo for Duodart plus lifestyle advice for 12 months
- Duodart: Participants received a combination of dutasteride 0.5 milligrams (mg) and tamsulosin 0.4 mg plus lifestyle advice for 12 months
Period: Overall Study
Arm/Group | Placebo | Duodart
Started | 246 | 243
Completed | 191 | 184
Not Completed | 55 | 59
Not completed — Adverse Event | 24 | 33
Not completed — Lack of Efficacy | 8 | 10
Not completed — Protocol Violation | 4 | 4
Not completed — Participants reached stopping criteria | 1 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 5 | 2
Not completed — Withdrawal by Subject | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Duodart: Participants received a combination of dutasteride 0.5 mg and tamsulosin 0.4 mg plus lifestyle advice for 12 months
- Total: Total of all reporting groups
Arm/Group | Placebo | Duodart | Total
Number analyzed (Participants) | 246 | 243 | 489
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (6.49) | 65.7 (6.59) | 65.5 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 246 | 243 | 489
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 2 | 3
  American Indian or Alaska Native | 2 | 3 | 5
  Asian - East Asian Heritage | 1 | 0 | 1
  White - Arabic/North African Heritage | 3 | 0 | 3
  White - White/Caucasian/European Heritage | 239 | 237 | 476
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline (BL) in Total Score From the Full Men's Sexual Health Questionnaire (MSHQ) at 12 Months
Description: Total MSHQ score is composed of 3 domain scores: Erection score(ES)=sum of score for Questions (Q) 1 to 3(ranges from 0 to 15), Ejaculation score(EjS)=sum of scores for Q5 to 11(ranges from 1 to 35), Satisfaction score(SS)=sum of scores for Q13 to 18(ranges from 6 to 30). Total MSHQ score=ES+EjS+SS. The total MSHQ score ranges from 7-80, with higher scores indicating greater sexual function. Change from BL at scheduled post-BL time points were analyzed using a mixed model repeated measures (MMRM) analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest double-blind (DB) treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 12 value(s) minus BL value(s)
Time Frame: Baseline and 12 months
Population: Intent-to-Treat (ITT): All randomized par. regardless of whether or not treatment was administered. Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 162 | 151
Scores on a scale | -0.7 (0.78) | -8.7 (0.81)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -8.00, 95% CI 2-sided [-10.22 to -5.79]

2. Secondary Outcome: Change From Baseline in Scores From the Full Men's Sexual Health Questionnaire (MSHQ) at 1, 3, 6 and 9 Months
Description: Total MSHQ score is composed of 3 domain scores: ES=sum of score for Q 1 to 3(ranges from 0 to 15), EjS=sum of scores for Q5 to 11(ranges from 1 to 35), SS=sum of scores for Q13 to 18(ranges from 6 to 30). Total MSHQ score=ES+EjS+SS and the score ranges from 7-80, with higher scores indicating greater sexual function. Change from BL at scheduled post-BL time points were analysed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 1, 3, 6, 9 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 1, 3, 6, and 9
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Month 1, n=193, 192 | -0.5 (0.68) | -4.6 (0.69)
  Month 3, n= 184, 181 | -0.5 (0.72) | -6.9 (0.73)
  Month 6, n=179, 164 | -0.8 (0.80) | -9.9 (0.83)
  Month 9, n=166, 146 | -0.8 (0.76) | -9.6 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -4.11, 95% CI 2-sided [-6.01 to -2.21] — Month 1
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, Adjusted mean difference; Adjusted mean difference = -6.43, 95% CI 2-sided [-8.45 to -4.41] — Month 3
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -9.04, 95% CI 2-sided [-11.31 to -6.77] — Month 6
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -8.82, 95% CI 2-sided [-10.96 to -6.67] — Month 9

3. Secondary Outcome: Number of Participants Reaching Various Thresholds of Change in Total MSHQ From Baseline at 12 Months
Description: Participants reaching thresholds of change in total MSHQ were assessed. Threshold values are defined as multiplicative factor. Threshold included +10 points, +20 points, +25 points, -10 points, -20 points, -25 points; where "+" indicates improvement and "-"indicates worsening. Treatment comparisons were done based on categories defined by these thresholds using Mantel-Haenszel test
Time Frame: Baseline and 12 months
Population: ITT Population; Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 162 | 151
Participants
  >= 25 | 0 | 1
  >= 20 | 3 | 3
  >= 10 | 16 | 8
  <= -25 | 3 | 13
  <= -20 | 3 | 20
  <= -10 | 24 | 61

4. Secondary Outcome: Change From Baseline in Erectile Dysfunction (ED) at 1, 3, 6, 9 and 12 Months
Description: Erection scale is a domain of MSHQ to assess erectile dysfunction. ES is the sum of score for questions 1 to 3. The score ranges from 0 (no erection) to 15 (strong erection). Change from BL at the scheduled post-baseline time points were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 1, 3, 6, 9 and 12 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 1, 3, 6, 9 and 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Month 1, n=209, 215 | -0.3 (0.15) | -0.5 (0.15)
  Month 3, n= 202, 208 | -0.5 (0.17) | -0.7 (0.17)
  Month 6, n= 193, 188 | -0.6 (0.18) | -1.0 (0.19)
  Month 9, n=182, 169 | -0.5 (0.18) | -1.2 (0.19)
  Month 12, n= 175, 168 | -0.5 (0.19) | -1.0 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.37, mixed-model repeated-measures; Adjusted mean difference = -0.20, 95% CI 2-sided [-0.62 to 0.23] — Month 1
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.33, mixed-model repeated-measures; Adjusted mean difference = -0.24, 95% CI 2-sided [-0.71 to 0.24] — Month 3
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.16, mixed-model repeated-measures; Adjusted mean difference = -0.37, 95% CI 2-sided [-0.88 to 0.15] — Month 6
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.009, mixed-model repeated-measures; Adjusted mean difference = -0.68, 95% CI 2-sided [-1.19 to -0.17] — Month 9
Statistical Analysis 5: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.091, mixed-model repeated-measures; Adjusted mean difference = -0.46, 95% CI 2-sided [-0.99 to 0.07] — Month 12

5. Secondary Outcome: Change From Baseline in Ejaculatory Dysfunction (EjD) at 1, 3, 6, 9 and 12 Months
Description: Ejaculation scale is a domain of MSHQ to assess ejaculatory dysfunction. EjS is the sum of score for questions 5 to 11. The score ranges from 1 (could not ejaculate) to 35 (strong ejaculation). Change from BL at the scheduled post-baseline time points were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 1, 3, 6, 9 and 12 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 1, 3, 6, 9 and 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Month 1, n=210, 208 | -0.3 (0.42) | -3.2 (0.43)
  Month 3, n= 197, 196 | -0.5 (0.48) | -5.8 (0.48)
  Month 6, n= 191, 179 | -0.7 (0.53) | -7.5 (0.54)
  Month 9, n=177, 161 | -0.5 (0.52) | -7.6 (0.53)
  Month 12, n= 173, 164 | -0.6 (0.55) | -7.5 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -2.89, 95% CI 2-sided [-4.07 to -1.70] — Month 1
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -5.24, 95% CI 2-sided [-6.59 to -3.90] — Month 3
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -6.82, 95% CI 2-sided [-8.30 to -5.34] — Month 6
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -7.05, 95% CI 2-sided [-8.51 to -5.59] — Month 9
Statistical Analysis 5: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -6.92, 95% CI 2-sided [-8.47 to -5.38] — Month 12

6. Secondary Outcome: Change From Baseline in Satisfaction Score at 1, 3, 6, 9 and 12 Months
Description: Satisfaction scale is a domain of MSHQ to assess sexual relationship. SS is the sum of score for questions 13 to 18. The score ranges from 6 (extremely dissatisfied) to 30 (extremely satisfied). Change from BL at the scheduled post-baseline time points were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 1, 3, 6, 9 and 12 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 1, 3, 6, 9 and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Month 1, n=200, 197 | 0.1 (0.26) | -0.8 (0.26)
  Month 3, n= 189, 182 | 0.4 (0.27) | -0.5 (0.28)
  Month 6, n= 185, 168 | 0.2 (0.30) | -1.5 (0.31)
  Month 9, n=173, 153 | -0.0 (0.30) | -1.2 (0.32)
  Month 12, n= 169, 152 | 0.3 (0.29) | -0.6 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.012, mixed-model repeated-measures; Adjusted mean difference = -0.94, 95% CI 2-sided [-1.67 to -0.21] — Month 1
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.017, mixed-model repeated-measures; Adjusted mean difference = -0.93, 95% CI 2-sided [-1.69 to -0.17] — Month 3
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -1.73, 95% CI 2-sided [-2.57 to -0.88] — Month 6
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.009, mixed-model repeated-measures; Adjusted mean difference = -1.15, 95% CI 2-sided [-2.01 to -0.30] — Month 9
Statistical Analysis 5: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.047, mixed-model repeated-measures; Adjusted mean difference = -0.83, 95% CI 2-sided [-1.65 to -0.01] — Month 12

7. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Scores Using the Observed Cases Approach at 2 Weeks, 1, 3, 6, 9, and 12 Months
Description: The IPSS questionnaire is a 7-item self-administered questionnaire designed to quantify urinary symptoms: Q1, incomplete emptying; Q2, frequency; Q3, intermittency; Q4, urgency; Q5, weak stream; Q6, straining; Q7, nocturia. The score can range from 0 to 35: mild (0 to 7), moderate (8 to 19), or severe (20 to 35). Change from BL were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Week 2, Months 1, 3, 6, 9 and 12 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 1, 3, 6, 9 and 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Week 2, n=232, 234 | -1.5 (0.29) | -3.1 (0.29)
  Month1, n=222, 231 | -2.8 (0.33) | -3.4 (0.33)
  Month 3, n=217, 224 | -2.8 (0.33) | -4.1 (0.33)
  Month 6, n=206, 203 | -2.9 (0.36) | -4.6 (0.36)
  Month 9, n=193, 185 | -3.2 (0.38) | -4.5 (0.38)
  Month 12, n=187, 184 | -3.2 (0.41) | -5.2 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -1.65, 95% CI 2-sided [-2.45 to -0.85] — Week 2
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.24, mixed-model repeated-measures; Adjusted mean difference = -0.55, 95% CI 2-sided [-1.47 to 0.37] — Month 1
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.006, mixed-model repeated-measures; Adjusted mean difference = -1.27, 95% CI 2-sided [-2.19 to -0.36] — Month 3
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -1.73, 95% CI 2-sided [-2.74 to -0.72] — Month 6
Statistical Analysis 5: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.013, mixed-model repeated-measures; Adjusted mean difference = -1.34, 95% CI 2-sided [-2.40 to -0.28] — Month 9
Statistical Analysis 6: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -1.97, 95% CI 2-sided [-3.12 to -0.83] — Month 12

8. Secondary Outcome: Change From Baseline in Quality of Life (BPH Impact Index -BII Scores) at 2 Weeks, 1, 3, 6, 9, and 12 Months
Description: The BPH Impact Index (BII) is a 4-item, self-administered questionnaire evaluating the impact of urinary problems on overall health and activity. Total scores range from 0 to 13; higher scores represent increased perceived impact of benign prostatic hyperplasia-lower urinary tract symptoms on overall health. Change from BL were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the subject took at least one dose of DB study drug; change from BL was calculated as Week 2, Months 1, 3, 6, 9 and 12 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 1, 3, 6, 9 and 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Week 2, n=226, 227 | -0.3 (0.14) | -0.7 (0.14)
  Month1, n=216, 223 | -0.7 (0.13) | -0.7 (0.13)
  Month 3, n=211, 217 | -0.9 (0.15) | -1.1 (0.15)
  Month 6, n=201, 195 | -0.6 (0.17) | -1.2 (0.17)
  Month 9, n=188, 179 | -0.7 (0.16) | -1.2 (0.17)
  Month 12, n=183, 177 | -0.6 (0.18) | -1.2 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.036, mixed-model repeated-measures; Adjusted mean difference = -0.40, 95% CI 2-sided [-0.78 to -0.03] — Week 2
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 1.00, mixed-model repeated-measures; Adjusted mean difference = 0.00, 95% CI 2-sided [-0.37 to 0.37] — Month 1
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.21, mixed-model repeated-measures; Adjusted mean difference = -0.26, 95% CI 2-sided [-0.67 to 0.15] — Month 3
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.009, mixed-model repeated-measures; Adjusted mean difference = -0.62, 95% CI 2-sided [-1.09 to -0.15] — Month 6
Statistical Analysis 5: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.056, mixed-model repeated-measures; Adjusted mean difference = -0.45, 95% CI 2-sided [-0.91 to 0.01] — Month 9
Statistical Analysis 6: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.023, mixed-model repeated-measures; Adjusted mean difference = -0.58, 95% CI 2-sided [-1.08 to -0.08] — Month 12

9. Secondary Outcome: Change From Baseline in Perception of Treatment Benefit/Satisfaction With Treatment (Patient Perception of Study Medication - PPSM Questionnaire Scores) at 2 Weeks, 1, 3, 6, 9, and 12 Months
Description: Patient Perception of Study Medication (PPSM) is a 12-item questionnaire designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms. The total PPSM score ranges from 7 to 49, with higher scores indicating lower satisfaction. Change from BL were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the subject took at least one dose of DB study drug; change from BL was calculated as Week 2, Months 1, 3, 6, 9, 12 values minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline, Week 2, Month 1, 3, 6, 9 and 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  Week 2, n=225, 227 | -0.4 (0.32) | -3.4 (0.32)
  Month1, n=216, 223 | -1.3 (0.38) | -3.4 (0.38)
  Month 3, n=211, 217 | -1.7 (0.41) | -3.8 (0.41)
  Month 6, n=201, 195 | -1.0 (0.44) | -3.6 (0.44)
  Month 9, n=188, 179 | -1.6 (0.45) | -2.9 (0.45)
  Month 12, n=182, 177 | -1.0 (0.49) | -4.6 (0.49)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -3.00, 95% CI 2-sided [-3.89 to -2.10] — Week 2
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -2.10, 95% CI 2-sided [-3.15 to -1.06] — Month 1
Statistical Analysis 3: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -2.11, 95% CI 2-sided [-3.25 to -0.98] — Month 3
Statistical Analysis 4: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -2.53, 95% CI 2-sided [-3.76 to -1.30] — Month 6
Statistical Analysis 5: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p = 0.042, mixed-model repeated-measures; Adjusted mean difference = -1.30, 95% CI 2-sided [-2.56 to -0.05] — Month 9
Statistical Analysis 6: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -3.51, 95% CI 2-sided [-4.87 to -2.14] — Month 12

10. Secondary Outcome: Change From Baseline in Total MSHQ Scores From Baseline at 12 Months Among Participants With IPSS Improvement of >=2 Points and >=3 Points
Description: Total MSHQ score is composed of 3 domain scores: ES+EjS+SS and the score ranges from 7-80, with higher scores indicating greater sexual function. Par. with change from baseline in total MSHQ scores with good BPH symptomatic response (measured by improvement in IPSS)were analysed. Change from BL at the scheduled post-baseline time points were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 12 value(s) minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 246 | 243
Scores on a scale
  IPSS improvement of >=2, n=152, 142 | -0.6 (0.81) | -8.4 (0.83)
  IPSS improvement of >=3, n=138,136 | -0.6 (0.86) | -8.0 (0.86)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -7.78, 95% CI 2-sided [-10.07 to -5.49] — Par. with IPSS change from baseline >=2 points improvement at any time post-baseline visit
Statistical Analysis 2: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -7.39, 95% CI 2-sided [-9.79 to -4.99] — Par. with IPSS change from baseline >=3 points improvement at any time post-baseline visit

11. Secondary Outcome: Change From Baseline in Total MSHQ Scores From Baseline at 12 Months Among Participants With IPSS Improvement of >=25 Percent
Description: Participants with change from baseline in total MSHQ scores with good BPH symptomatic response (measured by improvement in IPSS)were analysed.Change from BL at the scheduled post-baseline time points were analyzed using MMRM analysis method with an Observed Cases approach. Values are expressed as adjusted mean along with standard error. The MMRM analysis included fixed categorical effects of treatment, visit and treatment by visit interaction and the continuous fixed covariates of BL total score and BL score by visit interaction. BL is defined as earliest DB treatment start date if the par. took at least one dose of DB study drug; change from BL was calculated as Month 12 value(s) minus BL value(s). Only those par with non-missing change from baseline data were analysed (presented as n=X,X in the category titles)
Time Frame: Baseline and Month 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Duodart
Number analyzed (Participants) | 139 | 133
Scores on a scale | -0.6 (0.86) | -8.3 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Duodart; Test type: Superiority or Other; p < 0.001, mixed-model repeated-measures; Adjusted mean difference = -7.79, 95% CI 2-sided [-10.22 to -5.35] — Par. with IPSS change from baseline >=25 points improvement at any time post-baseline visit

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious Adverse Events (AEs) were collected from the start of study medication until follow-up (up to approximately 18 months).
Description: On-treatment SAEs and non-serious AEs are reported for ITT Population.
Arm/Group | Placebo | Duodart
Serious Adverse Events (participants affected / at risk) | 9/246 | 27/243
Other Adverse Events (participants affected / at risk) | 28/246 | 66/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=246) | Duodart (N=243)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fistula (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=246) | Duodart (N=243)
Erectile dysfunction (Reproductive system and breast disorders) | 16 (17) | 24 (25)
Retrograde ejaculation (Reproductive system and breast disorders) | 3 (3) | 23 (23)
Ejaculation disorder (Reproductive system and breast disorders) | 2 (2) | 16 (16)
Libido decreased (Psychiatric disorders) | 12 (12) | 20 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.